CLINICAL TRIAL: NCT00692432
Title: Macrophage Inhibitory Factor (MIF) and High-Mobility Group-1 Protein (HMG-1) in Children Undergoing Cardiopulmonary Bypass
Brief Title: Macrophage Inhibitory Factor and High-Mobility Group-1 Protein in Children Undergoing Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Children's Medical Center Dallas (Other)
Responsible Party: Principal Investigator, Leslie Garner, Assistant Professor of Pediatrics, University of Texas Southwestern Medical Center
Other Study IDs: 0901-475
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Myocardial Depression
Keywords: Macrophage Migration Inhibitory Factor; MIF; Cardiopulmonary bypass; CPB; inflammation; inflammatory marker; myocardial depression; myocardial depressant factor
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cardiac tissue serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Introduction: In recent scientific literature, 2 proteins, macrophage migration inhibitory factor (MIF) and high-mobility group-1 protein (HMG-1), have emerged as important mediators of inflammation and sepsis.

Hypothesis: MIF and HMG-1 will be present in the serum of children who have undergone cardiopulmonary bypass. MIF will be present in the myocardium of children who have undergone cardiopulmonary bypass. The presence of MIF and HMG-1 in the serum and MIF in the myocardium of children undergoing bypass will correlate with clinical outcome.

Methods: We will study a group of infants and children undergoing operative repair of congenital heart disease during which there is an expectation of cardiac tissue removal. Patients will have an assessment of cardiac function by echocardiography as well as blood assays for tumor necrosis factor (TNF), interleukin-6, interleukin-8, interleukin-10, MIF, and HMG-1 prior to surgery. Cardiac tissue, removed as a planned part of the procedure, will be obtained from the cardiothoracic surgeons and assayed for MIF and for apoptosis, a potential mechanism of myocardial dysfunction mediated by MIF and/or HMG-1. The patient will be admitted to the cardiac intensive care unit post operatively for routine care. Blood will be obtained at 1, 8, 24, 28, and 72 hours post operatively for the cytokine assays detailed above. The blood will be drawn from indwelling arterial or venous catheters routinely placed at the time of surgery. The amount of blood drawn (-4cc per sample) is unlikely to cause any hemodynamic compromise or result in additional blood product replacement.

Sample size and Analysis Plan: 30 subjects will be enrolled to determine the presence or absence of MIF/HMG-1 in the serum and cardiac tissue pre and post cardiopulmonary bypass. Descriptive statistics of patient demographics and clinical outcome variables will be correlated to serum and myocardial concentrations of the various cytokines.

DETAILED DESCRIPTION:
PURPOSE: To document the presence or absence of the proinflammatory cytokines macrophage migration inhibitory factor (MIF) and high-mobility group-1 protein (HMG-1) in the serum and myocardium of children undergoing cardiopulmonary bypass (CPB) and to correlate the presence or absence of these cytokines with clinical outcome after CPB

BACKGROUND: MIF, a 12.5 kD protein discovered in the 1960s as a substance produced by sensitized T lymphocytes involved in delayed type hypersensitivity, has emerged as a key cytokine in the innate immune response to infectious and inflammatory stimuli. Sources of MIF include monocytes/macrophages, the anterior pituitary, liver, kidney, spleen, and brain. MIF is released in response to various stimuli including lipopolysaccharide (LPS), toxic shock syndrome toxin-1, tumor necrosis factor (TNF), and interferon (INF). Once released, MIF promotes the secretion of other proinflammatory mediators by macrophages and T-cells thus intensifying the body's immune response. In addition, MIF has the unique ability to override the anti-inflammatory and immunosuppressive effects of glucocorticoids (Calandra et al., Nature Medicine, Feb 2000). MIF in combination with LPS potentiates lethality in murine endotoxemia models, and administration of anti-MIF antibodies increases survival in murine sepsis models. (Calandra et al., Nature Medicine, Feb 2000). Additionally, MIF knockout mouse models are resistant to lethal doses of LPS (Bozza et al., J Exp Med, Jan 1999).

HMG-1, a 30kD protein discovered in 1973, is a nonhistone chromatin-associated protein that serves as a DNA binding protein involved in nucleosome stabilization, facilitation of gene transcription, and as a modulator of steroid home receptor activity. More recently HMG-1 has been implicated as a monocyte/macrophage derived cytokine that serves as a late mediator of endotoxin lethality (Wang et al., Science 1999). Murine and human macrophages/monocytes release large amounts of HMG-1 18 hours after exposure to bacterial endotoxin. Serum HMG-1 levels rise 16-36 hours after LPS administration in murine lethal endotoxemia models. Administration of anti-HMG antibodies attenuates lethality in these models even when administered 2 hours after LPS exposure. Purified rHMG-1 is lethal to LPS-responsive and LPS-resistant mice. HMG-1 levels are increased in patients with sepsis and are higher in non-survivors than survivors. (Wang et al., Science 1999). HMG levels are also increased in patients with hemorrhagic shock (Ombrellino et al., Lancet 1999). HMG-1 induces TNF release by cultured human peripheral blood monocytes (Andersson et al., J Exp Med, 2000).

Cardiopulmonary bypass (CPB) triggers an inflammatory state associated with endotoxemia and cytokine elevation (Lequier et al., Chest, Jun 2000). Cytokines are known to have profound effects on cardiac function in sepsis. Cardiac depression occurs commonly after CPB and may be related to cytokine elevation. The role of MIF and HMG-1 in the CPB-induced inflammatory state are unknown. We have demonstrated the presence of MIF in murine heart tissue in response to LPS and are currently performing time course studies and functional assays examining murine cardiac myocyte response to MIF stimulus. In order to examine the clinical relevance of our laboratory data and to further characterize the inflammatory state occurring after CPB, we would like to obtain human data correlating MIF levels in human serum and myocardium with clinical outcome following CPB. Additionally, since the myocardial depression seen after CPB occurs 12-24 hours after CPB suggesting that a late mediator of inflammation may be important in post-CPB myocardial depression, we would like to assess for HMG-1 in the serum of patients undergoing CPB and correlate the presence or absence of HMG-1 with clinical outcome.

CONCISE SUMMARY OF PROJECT: We propose to study a population of infants and children undergoing operative repair of congenital heart disease during which there is an expectation that cardiac tissue will be removed. Patients will have an assessment of cardiac function by echocardiography as well as blood assays for tumor necrosis factor (TNF), interleukin-6, interleukin-8, interleukin-10, complement 3a, MIF, and HMG-1 prior to surgery. Cardiac tissue, removed as a planned part of the surgical procedure will be assayed for MIF as well as for evidence of apoptosis, a potential mechanism of cell death and myocardial dysfunction in response to MIF or HMG-1. The patients will be monitored in the PICU for a number of clinical outcome indicators including vital signs, fluid status, inotropic requirement, acid-base status, etc. Blood will be obtained prior to surgery and at 1, 8, 24, 48, and 72 hours post-operatively for cytokine assays to characterize the inflammatory response of each patient. We will then determine if MIF and/or HMG-1 levels correlate with clinical outcome.

SOURCES OF RESEARCH MATERIAL: Blood will be obtained pre- and postoperatively as described. Heart tissue will be obtained at the time of surgery as a routine part of the procedure. The biochemical assays performed on the samples are for research purposes only. Clinical data will be obtained from routinely recorded data from each patient's electronic PICU chart.

RECRIUTMENT OF SUBJECTS: Subjects will be recruited preoperatively in the cardiology clinic or PICU. Written informed consent will be obtained from a parent/legal guardian by one of the study investigators.

POTENTIAL RISKS: Study participation will not pose any additional discomfort or stress to the patient/family. Cardiac tissue removal will be a planned portion of the cardiac surgical repair regardless of study participation. Blood samples will be obtained from an indwelling vascular catheter routinely placed prior to surgery and will be collected at times when routine pre and post-operative tests are normally obtained. The amount of blood drawn (~4cc/sample) should not cause any hemodynamic compromise or result in additional blood product replacement. All patients will receive the same quality care and monitoring in the PICU regardless of study participation. Patients will not be responsible for any costs generated solely from research.

SPECIAL PRECAUTIONS: All blood samples will be obtained in a sterile fashion. Cardiac tissue will be obtained in the operating room as a routine part of the surgical procedure.

BIOSTATISTICS: A random sample of 30 subjects will be selected to determine whether or not MIF and HMG-1 are present in the cardiac tissue as well as serum obtained prior to and following CPB as outlined above. Descriptive statistics of patient demographics and plasma and tissue concentrations of indicated cytokines will be correlated to clinical outcome variables.

ELIGIBILITY:
Inclusion Criteria:

1. Any child under the age of 5 undergoing operative repair of congenital heart disease on CPB where there is an expectation of cardiac tissue removal.
2. Written informed consent obtained from a parent/legal guardian.

Exclusion Criteria:

1. Unable to obtain informed consent
2. Evidence of ongoing infection
3. Known immunodeficiency

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children at Children's Medical Center Dallas who are having cardiac surgery that requires CPB and an expectation of cardiac tissue removal.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2001-09; Primary Completion 2003-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
MIF and HMG-1 will be present in the serum of children who have undergone cardiopulmonary bypass. MIF will be present in the myocardium of children who have undergone cardiopulmonary bypass. | 72 hours

SECONDARY OUTCOMES:
MIF levels in human serum and myocardial cells will correlate with clinical outcome following CPB. | 72 hours
Presence or absence of HMG-1 in the serum of patients undergoing CPB will correlate with clinical outcome. | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Garner, MD, Principal Investigator — UT Southwestern
Locations (1):
- Children's Medical Center Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No